CLINICAL TRIAL: NCT00818753
Title: The Safety and Pharmacodynamics of Two Doses of Dabigatran Etexilate in Patients Undergoing Cardiac Catheterization
Brief Title: Randomized, Open Label Study of Dabigatran Etexilate in Elective Percutaneous Coronary Intervention
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1160.73; 2007-007536-25 (EudraCT Number: EudraCT)
Record Dates: First submitted 2009-01-07; First posted 2009-01-08 (Estimated); Results first posted 2011-10-25 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2013-12

CONDITIONS: Heart Catheterization
MeSH Terms: interventions — Dabigatran; Heparin

ARMS (3):
- Dabigatran 110 mg (Experimental): experimental drug therapy in this indication
  Interventions: Drug: dabigatran 110 mg
- Dabigatran 150 mg (Experimental): experimental drug therapy in this indication
  Interventions: Drug: dabigatran 150 mg
- Unfractionated Heparin (Active Comparator): standard therapy in this indication as comparator
  Interventions: Drug: unfractionated heparin

INTERVENTIONS:
Drug: dabigatran 110 mg — comparison of different dabigatran dosages with unfractionated heparin
  Arms: Dabigatran 110 mg
Drug: dabigatran 150 mg — comparison of different dabigatran dosages with unfractionated heparin
  Arms: Dabigatran 150 mg
Drug: unfractionated heparin — comparison of different dosages dabigatran with unfractionated heparin
  Arms: Unfractionated Heparin

SUMMARY:
To assess whether two doses of dabigatran etexilate (110 mg twice daily (b.i.d) and 150 mg twice daily (b.i.d)) as compared to unfractionated heparin (UFH), both in addition to a standard dual antiplatelet regimen, provide sufficient anticoagulation in the setting of elective percutaneous coronary intervention (PCI).

ELIGIBILITY:
Inclusion criteria:

* patients between 18 and 85 years
* due to undergo elective PCI
* informed consent obtained

Exclusion criteria:

* PCI lesion specific conditions
* class III or IV congestive heart failure
* severe hypertension
* increased bleeding risk
* thrombolytic therapy within 24 hours preceding randomization

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2009-01; Primary Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (4):
- Netherlands (4):
  - 1160.73.31004 Boehringer Ingelheim Investigational Site, Alkmaar
  - 1160.73.31003 Boehringer Ingelheim Investigational Site, Nieuwegein
  - 1160.73.1 Boehringer Ingelheim Investigational Site, Rotterdam
  - 1160.73.31002 Boehringer Ingelheim Investigational Site, Rotterdam

REFERENCES:
- [Derived] Vranckx P, Verheugt FW, de Maat MP, Ulmans VA, Regar E, Smits P, ten Berg JM, Lindeboom W, Jones RL, Friedman J, Reilly P, Leebeek FW. A randomised study of dabigatran in elective percutaneous coronary intervention in stable coronary artery disease patients. EuroIntervention. 2013 Jan 22;8(9):1052-60. doi: 10.4244/EIJV8I9A162. PMID 23182947

RESULTS

PARTICIPANT FLOW:
Groups:
- Heparin: Unfractionated heparin administered during intervention
Period: Overall Study
Arm/Group | Dabigatran 110mg Bis in Die (BID) | Dabigatran 150mg Bis in Die (BID) | Heparin
Started | 22 (There were 53 participants randomised, but only 51 were treated.) | 21 (There were 53 participants randomised, but only 51 were treated.) | 10 (There were 53 participants randomised, but only 51 were treated.)
Completed | 19 | 21 | 9
Not Completed | 3 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Other reason (not specified) | 0 | 0 | 1
Not completed — Randomised and not treated | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dabigatran 110mg Bis in Die (BID) | Dabigatran 150mg Bis in Die (BID) | Heparin | Total
Number analyzed (Participants) | 22 | 21 | 10 | 53
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.5 (8.7) | 63.0 (8.5) | 67.0 (8.3) | 64.8 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 3 | 17
  Male | 14 | 15 | 7 | 36
Race/Ethnicity, Customized [Number; unit: participants] — All participants were white
  participants | 22 | 21 | 10 | 53
Creatinine clearance [Mean (Standard Deviation); unit: mL/min] — Baseline creatinine clearance was not available for 3 patients in the Dabigatran 110mg treatment group.
  mL/min | 98.5 (38.2) | 96.3 (19.3) | 95.7 (26.5) | 97.0 (28.6)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Require Anticoagulation and/or Have Clinical Signs of Catheter Related Thrombosis
Description: Investigator reported outcome
Time Frame: From 22 to 165 minutes
Population: Full analysis set (FAS). All patients who were treated with randomised medication and underwent a cardiac intervention
Measure: Number; unit: Percentage of participants
Arm/Group | Dabigatran 110mg Bis in Die (BID) | Dabigatran 150mg Bis in Die (BID) | Heparin
Number analyzed (Participants) | 19 | 21 | 10
Percentage of participants | 10.5 (10.5) | 14.3 (14.3) | 10.0 (10)
Statistical Analysis 1: Comparison: Dabigatran 110mg Bis in Die (BID) vs Heparin; Dabigatran 110mg BID vs Heparin; Test type: Superiority or Other; Cochran-Mantel-Haenszel — p-values were not presented as the study was exploratory and not powered to to detect a difference in the treatments; Odds Ratio (OR) = 1.00, 95% CI [0.08 to 12.76]
Statistical Analysis 2: Comparison: Dabigatran 150mg Bis in Die (BID) vs Heparin; Dabigatran 150mg BID vs Heparin; Test type: Superiority or Other; Cochran-Mantel-Haenszel — p-values were not presented as the study was exploratory and not powered to to detect a difference in the treatments; Odds Ratio (OR) = 1.50, 95% CI [0.13 to 16.82]

2. Secondary Outcome: Percentage of Participants Who Experienced Catheter Related Thrombi Requiring Rescue Anticoagulation Therapy
Description: Investigator reported outcome
Time Frame: From 22 to 165 minutes
Population: Full analysis set. All patients who were treated with randomised medication and underwent a cardiac intervention
Measure: Number; unit: Percentage of participants
Arm/Group | Dabigatran 110mg Bis in Die (BID) | Dabigatran 150mg Bis in Die (BID) | Heparin
Number analyzed (Participants) | 19 | 21 | 10
Percentage of participants | 0 (0) | 0 (0) | 0 (0)

3. Secondary Outcome: Percentage of Participants Who Experienced Abrupt Vessel Closure, New Thrombus With Reduced Reflow or no Reflow
Description: Investigator reported outcome
Time Frame: From 22 to 165 minutes
Population: Full analysis set. All patients who were treated with randomised medication and underwent a cardiac intervention
Measure: Number; unit: Percentage of participants
Arm/Group | Dabigatran 110mg Bis in Die (BID) | Dabigatran 150mg Bis in Die (BID) | Heparin
Number analyzed (Participants) | 19 | 21 | 10
Percentage of participants | 10.5 (2) | 4.8 (1) | 0 (0)

4. Secondary Outcome: Percentage of Participants Who Experienced Catheter Related Thrombi Not Resulting in Clinical Complications Including Guide-catheter (Wire) Thrombosis
Description: Investigator reported outcome
Time Frame: From 22 to 165 minutes
Population: Full analysis set. All patients who were treated with randomised medication and underwent a cardiac intervention
Measure: Number; unit: Percentage of participants
Arm/Group | Dabigatran 110mg Bis in Die (BID) | Dabigatran 150mg Bis in Die (BID) | Heparin
Number analyzed (Participants) | 19 | 21 | 10
Percentage of participants | 0 (0) | 0 (0) | 0 (0)

5. Secondary Outcome: Number of Participants With Bleeding Events
Description: Bleeding is categorized using the TIMI criteria as major or minor bleeding. The time window for inclusion of bleeding events was up until 3 days post-procedure or discharge (whichever occurred first).
Time Frame: First administration until 7-14 days after PCI (Percutaneous Coronary Intervention)
Population: Treated set. All randomised patients who were documented to have taken at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Dabigatran 110mg Bis in Die (BID) | Dabigatran 150mg Bis in Die (BID) | Heparin
Number analyzed (Participants) | 20 | 21 | 10
participants | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: First administration until 7-14 days after PCI (Percutaneous Coronary Intervention)
Arm/Group | Dabigatran 110mg Bis in Die (BID) | Dabigatran 150mg Bis in Die (BID) | Heparin
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/21 | 0/10
Other Adverse Events (participants affected / at risk) | 4/20 | 3/21 | 3/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran 110mg Bis in Die (BID) (N=20) | Dabigatran 150mg Bis in Die (BID) (N=21) | Heparin (N=10)
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran 110mg Bis in Die (BID) (N=20) | Dabigatran 150mg Bis in Die (BID) (N=21) | Heparin (N=10)
Myocardial infarction (Cardiac disorders) | 1 | 2 | 0
Feeling cold (General disorders) | 1 | 1 | 0
Coronary artery occulsion (Cardiac disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
Ischaemia (Vascular disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Postinfaction angina (Cardiac disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Puncture site haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Although a total of 50 patients are included in the FAS, 4 of these patients did not have data for the primary endpoint and are therefore not included in the odd ratio calculation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.